CLINICAL TRIAL: NCT05560386
Title: TEEN HEED: An Adolescent Diabetes Prevention Intervention Incorporating Novel Mobile Health Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nita Vangeepuram, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 17-2272; 5R03DK118302-02 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12-16

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Text messaging program (Experimental): Enrolled participants received the pilot text messaging program.
  Interventions: Behavioral: Text messaging
- Virtual peer education (Experimental): Enrolled participants received a virtual peer education diabetes prevention program.
  Interventions: Behavioral: Virtual workshop

INTERVENTIONS:
Behavioral: Text messaging — text messaging content to support diabetes prevention.
  Arms: Text messaging program
Behavioral: Virtual workshop — virtual workshop content to support diabetes prevention.
  Arms: Virtual peer education

SUMMARY:
The number of youth with type 2 diabetes in the U.S. is projected to increase by a staggering 49 percent by 2050, with higher rates among minority youth. The Diabetes Prevention Program (DPP) is recognized as a sentinel study demonstrating the effectiveness of lifestyle interventions for diabetes prevention among pre-diabetic adults but has not yet been replicated in youth. In addition, such intensive interventions are often not sustainable in high risk communities with limited resources. One strategy that has been successfully employed in adults from such communities is peer based health education. However, there have been no peer led interventions in ethnic minority teens and no interventions focused specifically on weight loss for diabetes prevention. Another challenge identified in existing youth health intervention programs is keeping youth engaged to enhance program participation and impact. One potential strategy is the use of mobile technologies (text messaging, mobile applications, social media) to support weight management programs, but to date use of such technologies has largely not been studied in youth. The Principal Investigator's NIH Mentored Patient-Oriented Research Career Development Award (K23) aimed to use CBPR to develop and pilot test a peer-led diabetes prevention intervention incorporating mobile health technologies for at-risk adolescents. Based on results of focus groups which explored strategies for using peer educators and mHealth tools as part of a group lifestyle change program, the researchers did not find existing tools with all the features and functionalities required by users. The investigators therefore began working with teen stakeholders to create a new text messaging platform to support participants as the teens complete the intervention. This R03 research proposal aims to bring together clinical, technology and community experts to further develop and evaluate the mobile health platform. This will provide important pilot data to refine and disseminate the intervention for a larger RCT to be tested in a future R01.

Specific Aims:

1. Synthesize real-time data and analytics and conduct user interface (UI) testing to refine and enhance features of the prototype text messaging platform.
2. Investigate the potential for the developed platform to be used as an adjunct to a group educational intervention by examining whether level of use, user satisfaction, and degree of engagement with the platforms modifies behavioral and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1 (user interface testing):

* Ages 13-19 years;
* English speaking with English or Spanish speaking parent/guardian;
* Affiliated with East Harlem.

For Aim 2 (virtual workshop):

* Ages 13-19 years;
* English speaking with English or Spanish speaking parent/guardian;
* Affiliated with East Harlem;
* Overweight/obese based on measured body mass index;
* prediabetic based on hemoglobin A1c

Exclusion Criteria:

- Medical or developmental conditions which would make it difficult to participate in a virtual group educational program

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nita Vangeepuram, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Messaging Program | Virtual Peer Education
Started | 13 | 41
Completed | 13 | 24
Not Completed | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Text Messaging Program: Enrolled participants received the pilot text messaging program. Text messaging: text messaging content to support diabetes prevention.
- Total: Total of all reporting groups
Arm/Group | Text Messaging Program | Virtual Peer Education | Total
Number analyzed (Participants) | 13 | 41 | 54
Age, Customized [Mean (Standard Deviation); unit: years]
  Age for each arm | 18.54 (1.94) | 14.73 (1.72) | 15.65 (2.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 31
  Male | 3 | 20 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 23 | 33
  Not Hispanic or Latino | 3 | 11 | 14
  Unknown or Not Reported | 0 | 7 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 3 | 11 | 14
  Race: Hispanic or Latino | 10 | 22 | 32
  Race: White | 0 | 0 | 0
  Race: More than one race | 0 | 1 | 1
  Race: Unknown or Not Reported | 0 | 7 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 41 | 54

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: Maintenance or reduction of BMI after completion of the virtual diabetes prevention program.
  BMI is a person's weight in kilograms divided by the square of height in meters. A high BMI can indicate high body fatness and may lead to health problems.
Time Frame: baseline
Population: Data was not collected for the Text Messaging Program. It was a pilot feasibility and acceptability arm and no clinical and behavioral outcomes were collected for this group.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 24
kg/m^2 |  | 32.95 (6.72)

2. Primary Outcome: Body Mass Index (BMI)
Description: as for outcome 1
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 15
kg/m^2 |  | 32.8 (7.26)

3. Secondary Outcome: Number of Participants Who Were Responsive to Interactive 2-way Messages
Description: Text Messaging Program - Number of participants who were responsive to interactive 2-way messages
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Program
Number analyzed (Participants) | 13
Participants | 11

4. Secondary Outcome: Number of Participants Who Were Engaged Every Week
Description: Text Messaging Program - Number of participants who initially consented to the study who were engaged every week
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Program
Number analyzed (Participants) | 13
Participants | 9

5. Secondary Outcome: Level of Engagement
Description: Text Messaging Program - Level of engagement as measured by responsiveness to 2-way interactive messages.
  Percent responding over the 12 weeks.
Time Frame: Over 12 weeks of time
Measure: Number; unit: percent
Arm/Group | Text Messaging Program
Number analyzed (Participants) | 13
percent
  0-10% of the time | 0
  11-25% of the time | 15
  26-50% of the time | 31
  51-75% of the time | 8
  >75% of the time | 46

6. Secondary Outcome: Hemoglobin A1c
Description: A1C is a lab test that shows the average level of blood sugar (glucose) over the previous 3 months. It shows how well a person is controlling blood sugar to help prevent complications from diabetes.
  Hemoglobin A1c (per American Diabetes Association): normal is 4-5.6% (5.7-6.4% is prediabetes and >6.5% is diabetes level)
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 25
percentage of red blood cells |  | 5.85 (0.20)

7. Secondary Outcome: Hemoglobin A1c
Description: as for outcome 6
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 12
percentage of red blood cells |  | 5.75 (0.20)

8. Secondary Outcome: Body Fat %
Description: For girls normal range is 16-31% for ages 13-18 years; for boys normal range is 10-22% for ages 13-18 years. Higher % indicates higher metabolic risk.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 18
percentage of fat |  | 37.27 (10.46)

9. Secondary Outcome: Body Fat %
Description: as for outcome 8
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
percentage of fat |  | 36.16 (8.27)

10. Secondary Outcome: Waist Circumference
Description: Waist circumference for boys/girls 10th-90th percentile ranges from 63.0-116.5 cm. Higher percentile indicates higher metabolic risk.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 18
cm |  | 103.01 (18.78)

11. Secondary Outcome: Waist Circumference
Description: as for outcome 10
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 15
cm |  | 104.45 (13.69)

12. Secondary Outcome: Blood Pressure - Systolic and Diastolic Blood Pressures
Description: Blood pressure is the pressure of circulating blood against the walls of blood vessels. Higher blood pressure may indicate higher metabolic risk.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 26
mmHg
  Systolic |  | 117.58 (6.47)
  Diastolic |  | 63.69 (6.78)

13. Secondary Outcome: Blood Pressure - Systolic and Diastolic Blood Pressures
Description: as for outcome 12
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 12
mmHg
  systolic |  | 115.33 (9.52)
  diastolic |  | 62.67 (6.30)

14. Secondary Outcome: Total Cholesterol
Description: (<200 is low risk, 200-239 borderline, >240 high risk).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 12
mg/dL |  | 175.83 (32.03)

15. Secondary Outcome: Total Cholesterol
Description: (<200 is low risk, 200-239 borderline, >240 high risk).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 4
mg/dL |  | 171.25 (36.23)

16. Secondary Outcome: Low Density Lipoprotein (LDL)
Description: (<100 is best, 100-129 is acceptable for those with no health issues, 130-159 is borderline, 160-189 is high).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 19
mg/dL |  | 97.85 (31.08)

17. Secondary Outcome: Low Density Lipoprotein (LDL)
Description: (<100 is best, 100-129 is acceptable for those with no health issues, 130-159 is borderline, 160-189 is high).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 7
mg/dL |  | 109.46 (39.37)

18. Secondary Outcome: High Density Lipoprotein (HDL)
Description: (>60 is good, 40-59 is normal, <40 is associated with increased risk of heart disease).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 21
mg/dL |  | 47.34 (21.14)

19. Secondary Outcome: High Density Lipoprotein (HDL)
Description: (>60 is good, 40-59 is normal, <40 is associated with increased risk of heart disease).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 7
mg/dL |  | 42.14 (7.93)

20. Secondary Outcome: Triglycerides
Description: (<150 is normal, 150-199 is borderline, 200-499 is high).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 15
mg/dL |  | 110.4 (78.29)

21. Secondary Outcome: Triglycerides
Description: (<150 is normal, 150-199 is borderline, 200-499 is high).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 4
mg/dL |  | 73.5 (42.13)

22. Secondary Outcome: Portion Control
Description: This is a validated scale to measure how well someone controls the amount of food they eat. The total scale value ranges from 8-32; higher score indicates better portion control.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 34
score on a scale |  | 22 (3.4)

23. Secondary Outcome: Portion Control
Description: as for outcome 22
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 25.1 (3.7)

24. Secondary Outcome: Self-Efficacy Healthy Eating Subscale 1
Description: This is a validated scale to measure how confident someone is that they can eat healthy. The total scale value ranges from 8-40; higher score indicates higher self-efficacy.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 24.8 (8)

25. Secondary Outcome: Self-Efficacy Healthy Eating Subscale 1
Description: as for outcome 24
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 26.9 (7.3)

26. Secondary Outcome: Self-Efficacy Health Eating Subscale 2
Description: This is a validated scale to measure how confident someone is that they can eat healthy. The total scale value ranges from 5-25; higher score indicates higher self-efficacy.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 18.7 (4.4)

27. Secondary Outcome: Self-Efficacy Health Eating Subscale 2
Description: as for outcome 26
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 18.9 (5.3)

28. Secondary Outcome: Perceived Barriers to Health Eating
Description: This is a scale to measure participants perceptions about the barriers they face for eating healthy. The total scale value ranges from 4-16; higher score indicates more perceived barriers.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 9.5 (2.1)

29. Secondary Outcome: Perceived Barriers to Health Eating
Description: as for outcome 28
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 7.7 (2.2)

30. Secondary Outcome: Daily MVPA Hours
Description: Daily MVPA (moderate to vigorous physical activity) hours of moderate to vigorous physical activity (daily, average over the last week)
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 1.1 (0.4)

31. Secondary Outcome: Daily MVPA Hours
Description: as for outcome 30
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 1.4 (0.4)

32. Secondary Outcome: Strenuous Exercise Hours
Description: Hours of strenuous physical activity (daily, average over the last week).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 0.5 (0.3)

33. Secondary Outcome: Strenuous Exercise Hours
Description: Hours of strenuous physical activity (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.7 (0.2)

34. Secondary Outcome: Moderate Exercise Hours
Description: Hours of moderate physical activity (daily, average over the last week).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 0.6 (0.3)

35. Secondary Outcome: Moderate Exercise Hours
Description: Hours of moderate physical activity (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.7 (0.2)

36. Secondary Outcome: Mild Exercise Hours
Description: Hours of mild physical activity (daily, average over the last week).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 0.6 (0.4)

37. Secondary Outcome: Mild Exercise Hours
Description: Hours of mild physical activity (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.7 (0.2)

38. Secondary Outcome: Time Spent Doing Physically Active Chores
Description: Hours of physically active chores (daily, average over the last week).
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Time Spent Doing Physically Active Chores
Description: Hours of physically active chores (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.8 (0.3)

40. Secondary Outcome: Time Spent Walking
Description: Hours of walking (daily, average over the last week).
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Time Spent Walking
Description: Hours of walking (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.7 (0.4)

42. Secondary Outcome: Time Spent Doing Unscheduled/Unstructured Physical Activity
Description: Hours of Unscheduled/unstructured PA (daily, average over the last week).
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Time Spent Doing Unscheduled/Unstructured Physical Activity
Description: Hours of Unscheduled/unstructured PA (daily, average over the last week).
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 0.7 (0.3)

44. Secondary Outcome: Screentime -Weekday
Description: Screen time on the weekdays in hours (daily, average) - Combined TV, computer, video games, smartphone/Ipad/etc.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 7.7 (3.2)

45. Secondary Outcome: Screentime -Weekday
Description: Screen time on the weekdays in hours (daily, average) - Combined TV, computer, video games, smartphone/Ipad/etc.
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 5.9 (2.3)

46. Secondary Outcome: Screentime-weekend
Description: Screen time on the weekend in hours (daily, average) - Combined TV, computer, video games, smartphone/Ipad/etc.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
hours |  | 17.3 (4.4)

47. Secondary Outcome: Screentime-weekend
Description: Screen time on the weekend in hours (daily, average) - Combined TV, computer, video games, smartphone/Ipad/etc.
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
hours |  | 15.6 (4.2)

48. Secondary Outcome: Physical Activity Self Efficacy Score
Description: This is a validated scale to measure how confident participants are that they can be physically active. The total scale value ranges from 6-24; higher score indicates higher self-efficacy.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 19.8 (5.6)

49. Secondary Outcome: Physical Activity Self Efficacy Score
Description: This is a validated scale to measure how confident participants are that they can eat healthy. The total scale value ranges from 6-24; higher score indicates higher self-efficacy.
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 13
score on a scale |  | 20.2 (5.5)

50. Secondary Outcome: Perceived Barriers to Physical Activity Score
Description: This is a scale to measure participants perceptions about the barriers they face for being physically active. The total scale value ranges from 8-32; higher score indicates more perceived barriers.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 15.4 (3.5)

51. Secondary Outcome: Perceived Barriers to Physical Activity Score
Description: This is a scale to measure participants perceptions about the barriers they face for eating healthy. The total scale value ranges from 8-32; higher score indicates more perceived barriers.
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 14.2 (3.8)

52. Secondary Outcome: Self-Image Score
Description: Total range score from 6-24; higher score indicates better self-image
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Self-Image Score
Description: Total range score from 6-24; higher score indicates better self-image
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 16.1 (3.3)

54. Secondary Outcome: Depression Score
Description: Total range score from 6-18; higher score indicates more depression symptoms
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Depression Score
Description: Total range score from 6-18; higher score indicates more depression symptoms
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 10.9 (3.5)

56. Secondary Outcome: Body Satisfaction Score
Description: Total range score from 10-60; higher score indicates higher body satisfaction
Time Frame: baseline
Population: This outcome was not included in the baseline survey.
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Body Satisfaction Score
Description: Total range score from 10-60; higher score indicates higher body satisfaction
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 27.1 (8.1)

58. Secondary Outcome: Emotional Eating Score
Description: Total range score from 5-20; higher score indicates more emotional eating
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 35
score on a scale |  | 8 (2.9)

59. Secondary Outcome: Emotional Eating Score
Description: Total range score from 5-20; higher score indicates more emotional eating
Time Frame: end of study at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Program | Virtual Peer Education
Number analyzed (Participants) | 0 | 14
score on a scale |  | 6.6 (2.1)

ADVERSE EVENTS:
Time Frame: end of study at 3 months
Arm/Group | Text Messaging Program | Virtual Peer Education
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/24
Other Adverse Events (participants affected / at risk) | 0/13 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05560386/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05560386/ICF_001.pdf